CLINICAL TRIAL: NCT05767502
Title: Investigation of the Effect of Assigning Verbal Component Score to Glasgow Coma Scale in Patients With Traumatic Brain Injury and Adding Pupil Reaction to Determining Mortality/Morbidity in Patients
Brief Title: Assignment of the Verbal Component Score and Addition of Pupil Reaction to the Glasgow Coma Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, AKİF BULUT, Principal Investigator, Uludag University
Other Study IDs: 2019-KAEK-140
Record Dates: First submitted 2023-02-28; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Brain Injuries, Traumatic
Keywords: GCS; GCS-Pupil score; Brain trauma; Consciousness
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: GCS-Pupil score — GCS+attributed verbal score- Step 1 to obtain pupillary score:
  * Patients with a motor (M) and eye-opening response (E) total score between 2 and 6 are assigned a verbal score of +1
  * Patients with an M+E score of 7 are assigned a verbal score of +2
  * Patients with an M+E score of 8-9 are assigned a verbal score of +4
  * Patients with an M+E score of 10 are assigned a verbal score of +5
  GCS+attributed verbal score- Step 2 to obtain the pupillary score:
  The total score is obtained by subtracting the pupil score from the score obtained in the 1st step. Pupil score is scored as follows;
  * 0 points if both pupils react to light,
  * 1 point if a pupil does not react to light and has anisocoria,
  * 2 points if both pupils do not react to light
  Other Names: GCS+attributed verbal score- Pupil score

SUMMARY:
In this study, it is aimed to determine the prognostic value of GCS-P and the GCS-P score, which is formed by assigning a verbal score, in patients with traumatic brain injury, where all parameters can be evaluated. In the model to be created, a new total score will be obtained with Motor score + Eye Response + assigned verbal Score-Pupil score and this score will be compared with GCS and GCS-Pupil score.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital due to traumatic brain injury,
* 18 years and older,
* who were alive at the time of admission,
* Patients whose GCS and pupil reactivity can be evaluated completely.

Exclusion Criteria:

* Younger than 18,
* Not alive at the time of admission,
* Patients whose GCS score and pupil reactivity are not correctly evaluated (facial trauma, past eye diseases or eye defects, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: When α: 0.05 β: 0.20 and the acceptable difference between models were selected as 10% using the G-Power program, the number of patients to be included in the study was determined as 199.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
MORTALITY | From admission to discharge, an average of 1 weeks
  Death of the patient while in the hospital
MORBIDTIY | From admission to discharge, an average of 1 weeks
  Patients with a Glasgow Outcome score of 2 and 3 (Each patient can get 1-5 points from the Glasgow Outcome score. A low score indicates a negative result.

SECONDARY OUTCOMES:
MORTALITY | 3 months after hospital discharge
  Death within 3 months after hospital discharge
MORBIDITY | 3 months after hospital discharge
  A Glaskow Coma Outcome Score of 2 and 3 at the end of 3 months after discharge from the hospital. (Each patient can get 1-5 points from the Glasgow Outcome score. A low score indicates a negative result)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing of study data is not allowed in our country.